CLINICAL TRIAL: NCT07017894
Title: Applying Breast Mask Containing Cabbage Leaves Extract to Relieve Breast Discomfort in Breastfeeding Women：A Double-blind Randomized Controlled Trial
Brief Title: Applying Breast Mask Containing Cabbage Leaves Extract to Relieve Breast Discomfort in Breastfeeding Women
Acronym: BMCCLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-04-009A; ACIC-114-005 (Other: Taipei Veterans General Hospital)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Breast Engorgement
Keywords: breast engorgement; pain; hardness
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: two-group pre-test and repeated post-test study design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breast mask containing cabbage leaves extract group (Experimental): Apply the breast mask containing cabbage leaf extract to the breasts, avoiding the nipples, for 20 minutes, 2 times a day, for 3 days.
  Interventions: Combination Product: Experimental: breast mask containing cabbage leaves extract group
- breast mask without cabbage leaves extract group (Sham Comparator): Apply a breast mask without cabbage leaves extract to the breasts, avoiding the nipples, for 20 minutes, 2 times a day, for 3 days.
  Interventions: Combination Product: Sham Comparator

INTERVENTIONS:
Combination Product: Experimental: breast mask containing cabbage leaves extract group — apply breast mask to the breasts, avoiding the nipples, for 20 minutes, 2 times a day, for 3 days
  Arms: breast mask containing cabbage leaves extract group
Combination Product: Sham Comparator — Apply a breast mask without cabbage leaves extract to the breasts, avoiding the nipples, for 20 minutes, 2 times a day, for 3 days.
  Arms: breast mask without cabbage leaves extract group

SUMMARY:
In this article, women were randomly assigned to the Breast Mask Containing Cabbage Leaves Extract group and Breast Mask without Cabbage Leaves Extract group, and the breast engorgement, pain, hardness, before and after each treatment were measured. At the end of the study breast mask user experience and continued breastfeeding were measured.

DETAILED DESCRIPTION:
Breast engorgement as the swelling and distention of breast, which is one of the most common problems often occurs 2-4 days after delivery, resulting in pain and fever, which reduces the intention of mothers to continue breastfeeding and causes to stop breastfeeding in the early postpartum period.

There are many conservative treatments for relieving breast engorgement. At present, there have been published studies on the application of medications, cold compresses, warm compresses, massages, gua sha and cabbage leaves compression to breast problems during lactation. Previous studies have shown that cabbage leaves compression can relieve the breast engorgement, pain, and hardness of postpartum women. However, safety concerns related to freshness, preservation, and residual pesticides must be considered when using cabbage leaves in a clinical setting. The purpose of this study was to examine whether breast mask containing cabbage leaves extract can improve breast engorgement, pain, and hardness.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Breastfeeding.
* Physiological breast swelling, breast heaviness, lumps, milk plugging, breast pain after childbirth.
* Able to read and understand Chinese.

Exclusion Criteria:

* Stillbirth
* Allergy to cabbage or sulfa.
* lactation inhibitors agents used.
* Fever symptoms (> 38 degrees Celsius), including: wound infection, upper respiratory tract infection, urinary tract infection.
* Breast symptoms, including: nipple cracks, skin damage, breast abscesses, mastitis, Malignant tumors.
* Postpartum complications, including: postpartum hemorrhage, amniotic fluid embolism or other diseases requiring close care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — yes
Enrollment: 154 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Breast engorgement_self-rating scale | Day1, 2, 3
  Total four items of breast engorgement, pain, hardness, and heat. There are eleven grades, a score of 0 represents no problem at all, and a score of 10 represents the most severe degree.
Breast hardness_Physiological measurements | Day1,2,3.
  NEUTONE TDM-Z2 durometer pressure gauge

SECONDARY OUTCOMES:
Breast mask user experience | Day 3
  Does Pleura fit your needs? Pleural comfort level? Purchase intention? Recommend others to buy? How much would you consider buying it at?
Continued breastfeeding | Day 30
  Total five items. There are five items of Exclusive breastfeeding/breastfeeding, Exclusive breastfeeding/bottle feeding, Exclusive breastfeeding/breastfeeding and bottle feeding, Mixed feeding, Feeding formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided